CLINICAL TRIAL: NCT06238063
Title: Implementing a Nurse-led Advance Care Planning (ACP) Intervention to Improve ACP Uptake in Residential Care Homes: An Implementation Science and Mixed Methods Pragmatic Cluster Randomized Controlled Trial
Brief Title: Implementing a Nurse-led Advance Care Planning (ACP) Intervention in Residential Care Homes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW 22-021
Record Dates: First submitted 2023-03-23; First posted 2024-02-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Advanced Care Planning
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The ACP intervention, which was developed by the expert panel, will be delivered by trained nurses in each RCH during a mandatory annual individual care planning (ICP) meeting. Eligible residents and their family members will be invited to attend the ICP meeting with ACP discussion.
  Interventions: Behavioral: Nurse-led Advance Care Planning (ACP) Intervention
- Control (No Intervention): Participants in the control arm will receive usual care with no ACP intervention.

INTERVENTIONS:
Behavioral: Nurse-led Advance Care Planning (ACP) Intervention — An ACP discussion between the participating resident, family members, and the trained nurse will be incorporated into the annual review. The proposed ACP intervention will be divided into three parts (three weekly sessions, 1.5 hours each): 1) preparatory, 2) discussion, and 3) follow-up sessions.
  Arms: Intervention

SUMMARY:
The goal of this cluster randomized controlled trial is to examine the effectiveness of a nurse-led advance care planning (ACP) intervention on improving ACP discussion uptake in residential care homes (RCHs). The main question it aims to answer is: The effectiveness of nurse-led advance care planning (ACP) interventions implemented on eligible residents in residential care homes on improving ACP discussion uptake in this population.

Compared to participants in the control group who will only receive usual care with no ACP intervention, residents and their family members in the intervention group will be invited to attend the ICP meeting with ACP discussion. The ACP discussion will be guided by the established protocol, which was developed by the expert panel and delivered by trained nurses.

DETAILED DESCRIPTION:
Targeted issue: The lack of ACP discussion and poor dyadic congruence pose challenges to the provision of good EOL care in Hong Kong RCHs.

Population: RCHs in Hong Kong with nurse-to-resident ratios ≥1:3 will be targeted to ensure adequate staffing to carry out ACP. Eligible participants have to be age 65 or older and be able to communicate in Cantonese or Mandarin. Participants will also be invited to identify family members involved in making decisions about their care to participate in the intervention.

Intervention: a nurse-led advance care planning (ACP) intervention

Main study aim: To implement a nurse-led ACP intervention for improving ACP uptake in RCH residents in Hong Kong to bridge the evidence-practice gap.

Study method: This implementation science study will use a mixed methods approach, including a pair-matched cluster-RCT and qualitative interviews, and relevant outcomes will be followed for up to 2 years. RCHs will be randomized into two groups: a nurse-led ACP intervention group and a control group with usual care only.The ACP documentation (i.e., new documentation related to ACP and EOL care) in medical records of all RCH residents in the intervention and control groups will be audited by the research team at baseline (T0), post-intervention (T1; after the ACP intervention), 1-year follow-up (T2; 1 year after the launch of the ACP intervention at the RCH), and 2-year follow-up (T3; 2 years after the launch of the ACP intervention at the RCH).

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants have to be age 65 or older and be able to communicate in Cantonese or Mandarin.
* Participants will also be invited to identify family members involved in making decisions about their care to participate in the intervention. For residents who have moderate or severe cognitive impairment (as determined by a score of less than 19 in the Hong Kong version of the Montreal Cognitive Assessment), the participation of family members is mandatory.

Exclusion Criteria:

* They have a moderate or severe significant cognitive impairment but do not have family members, or
* They have prior ACP experience (e.g., AD completed).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Chart review at post-intervention | baseline and immediately after the intervention
  The medical records of all RCH residents will be audited at baseline (T0), post-intervention (T1; after the ACP intervention), 1-year follow-up (T2; 1 year after the launch of the ACP intervention at the RCH), and 2-year follow-up (T3; 2 years after the launch of the ACP intervention at the RCH). The following information will be extracted: ACP documentation (primary outcome; i.e., new documentation related to ACP and EOL care); designated surrogate decision-maker; AD completion; and healthcare utilization (i.e., number of inpatient hospitalizations, emergency department visits, intensive care unit admissions and length of stay, mechanical intubation rates and in-hospital cardiopulmonary resuscitation rates during the 6 months before death, place of death). The information specific to ACP intervention will only be extracted in residents who participated in ACP intervention: concordance on EOL preferences ; and concordance between preferred and actual outcomes of EOL care.
Change from Baseline in Chart review at 1-year follow-up time point. | 1-year follow-up (i.e., 1 year after the launch of the ACP intervention)
  The medical records of all RCH residents will be audited at baseline (T0), post-intervention (T1; after the ACP intervention), 1-year follow-up (T2; 1 year after the launch of the ACP intervention at the RCH), and 2-year follow-up (T3; 2 years after the launch of the ACP intervention at the RCH). The following information will be extracted: ACP documentation (primary outcome; i.e., new documentation related to ACP and EOL care); designated surrogate decision-maker; AD completion; and healthcare utilization (i.e., number of inpatient hospitalizations, emergency department visits, intensive care unit admissions and length of stay, mechanical intubation rates and in-hospital cardiopulmonary resuscitation rates during the 6 months before death, place of death). The information specific to ACP intervention will only be extracted in residents who participated in ACP intervention: concordance on EOL preferences ; and concordance between preferred and actual outcomes of EOL care.
Change from Baseline in Chart review at 2-year follow-up time point. | 2-year follow-up (i.e., 2 years after the launch of the ACP intervention at the RCH).
  The medical records of all RCH residents will be audited at baseline (T0), post-intervention (T1; after the ACP intervention), 1-year follow-up (T2; 1 year after the launch of the ACP intervention at the RCH), and 2-year follow-up (T3; 2 years after the launch of the ACP intervention at the RCH). The following information will be extracted: ACP documentation (primary outcome; i.e., new documentation related to ACP and EOL care); designated surrogate decision-maker; AD completion; and healthcare utilization (i.e., number of inpatient hospitalizations, emergency department visits, intensive care unit admissions and length of stay, mechanical intubation rates and in-hospital cardiopulmonary resuscitation rates during the 6 months before death, place of death). The information specific to ACP intervention will only be extracted in residents who participated in ACP intervention: concordance on EOL preferences ; and concordance between preferred and actual outcomes of EOL care.

OTHER OUTCOMES:
Quality about End-of-life Communication (QOC) | immediately after the intervention and 2 years after the launch of intervention.
  ACP discussion quality will be assessed by the QOC questionnaire, a 13-item instrument that consists of an overall score and two subscale scores for "general communication skills" and "communication about end-of-life care".Residents and family member(s) that have participated in the ACP intervention will be invited to complete the questionnaire at at post-intervention and 2 years after the launch of the ACP intervention.
Caregiver quality-of-life (QOL) | baseline, immediately after the intervention, and 2 years after the launch of intervention.
  Informal caregivers' QOL will be assessed by the Quality of Life in Life Threatening Illness--Family Carer Version (QOLLTI-F), a 16-item instrument with seven subscales for state of carer, patient wellbeing, quality of care, outlook, environment, finances, and relationships. Family members participating in the ACP intervention will be invited to completed the questionnaire at baseline (T0), post-intervention (T1), and 2 years after the launch of intervention (T3).
Qualitative interviews | immediately after the intervention and 1 year after the launch of intervention
  Individual semi-structured interviews will be held at post-intervention (T1) and 1 year after the launch of intervention (T2) with residents and family members (regarding their experience of receiving the intervention) and 2) care homes managers and trained nurses (regarding their experience of delivering the intervention), and allied healthcare workers (including patient care assistants, social workers, and physiotherapists). 20 participants in each group will be invited for interviews. A purposive sampling method will be used with consideration of characteristics of participants and the residential care homes (e.g., high or low rates of ACP completion). Through the interviews, we aim to obtain in-depth understanding of their experience of receiving/implementing the ACP intervention. This approach will enhance the quality of the evaluation of implementation intervention effectiveness and provide insight into further improvements.
Recruitment data | baseline and 2 years after the launch of intervention
  The following outcomes will be calculated from the screening and recruitment data: eligibility rate (i.e., the proportion of residents in the intervention group eligible for the study); participation rate (i.e., the proportion of the eligible residents consenting to participant); sample representativeness (i.e., characteristics of residents engaged compared with all eligible residents); organizational adoption (i.e., percentage of RCHs where intervention was intended to be implemented that actually adopted the intervention); and provider adoption (i.e., number and proportion of nurses that attended training and initiated ACP intervention in real practice).
intervention fidelity | immediately after the intervention
  At post-intervention (T1), the intervention group nurses will complete the pre-designed fidelity checklist to assess the intervention fidelity, i.e., the extent to which the intervention components are delivered as planned.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chin Lin, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang T, Cheung DST, Chu C, Chen J, Lin CC. Evaluation of a train-the-trainer implementation strategy on providers' competency, opportunity and motivation for advance care planning in residential care homes: a mixed-methods study. BMC Geriatr. 2026 Jan 3. doi: 10.1186/s12877-025-06898-2. Online ahead of print. PMID 41484702